CLINICAL TRIAL: NCT03227107
Title: IRF-1 Regulate Alveolar Macrophage Pyroptosis in Acute Lung Injury and of Which Will be Possible Mechanism
Brief Title: The Evaluation of NETs, Caspase-1 and Cytokines in ARDS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, panpinhua, vice director of department of respiratory, Xiangya Hospital of Central South University
Other Study IDs: 81470266
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. enrollment criteria and clinical data collection: follow the principles of medical ethics, the development of inclusion and exclusion criteria, select 90 cases of ARDS patients, in the active treatment at the same time, according to the Berlin standard severity of the disease divided into mild group, moderate Group and severe group, according to the prognosis during hospitalization is divided into survival group and death group. BALF specimens were collected on the day of admission to detect the levels of NETs and alveolar macrophages. The acute and chronic health status scoring system Ⅱ (APACHEⅡ) and Murray acute lung injury score, blood routine, creatinine, urea nitrogen, fasting blood glucose, Item, mean arterial pressure, arterial blood gas analysis, oxygenation index; record the patient's mechanical ventilation time and other data;
2. Pearson linear correlation analysis of BALF in the content of NETs, alveolar macrophage coke death level was a positive correlation between the Spearman rank correlation analysis BALF in the NETs content and alveolar macrophage coke death level, APACHE Ⅱ, Murray score, creatinine, Urea nitrogen, fasting blood glucose and other indicators and ARDS severity was positively correlated;
3. To analyze the prognostic factors of different prognostic factors, to evaluate the content of NETs in BALF, the level of alveolar macrophage coke, APACHEⅡ and Murray scores were analyzed by receiver operator characteristic curve (ROC curve) Short - term survival outcome prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients diagnosis within 3 days
* Over 18 years old but no more than 75 years old

Exclusion Criteria:

* Severe thoracic open trauma
* Pulmonary embolism
* Severe cardiovascular and cerebrovascular disease
* Endocrine system diseases
* Coagulation dysfunction
* Liver and kidney failure
* Malignant tumors
* Cardiogenic pulmonary edema

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ARDS
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
neutrophil extracellular traps, caspase-1,cytokines measurement | 4 years
  Assessments with neutrophil extracellular traps be presented in ng/ml; Assessments with caspase-1 and cytokines be presented in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided